## **Study Title**

Double Blind Clinical Evaluation on the combination of Gamma-Aminobutyric Acid Tartrate 100mg, Glutamic Acid 100mg, Dibasic Calcium Phosphate 50mg, Thiamine Nitrate 25mg, Pyridoxine Hydrochloride 10mg and Cyanocobalamin 5mcg compared to Ginger Extract as adjuvant therapy in symptomatic control of chronic vertigo motion sickness

Study sample was estimated using Power & Precision software (version 4.0), upon the null hypothesis that the proportion of patients expected to show clinical improvement shall be the same between both study groups. Statistical significance level (alfa) was set as 0.05 and study test as two tailed. Study power is 36.4% in order to generate a statistical significant result assuming a population of 167 patients per group, with an estimated proportional difference between groups as 0.05.